CLINICAL TRIAL: NCT02363803
Title: Predicting Individual Response to Analgesic Treatment in Painful Diabetic Neuropathy
Brief Title: Lidocaine for Diabetic Peripheral Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, simon.haroutounian, Assistant Professor, Washington University School of Medicine
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 201412073
Record Dates: First submitted 2015-02-03; First posted 2015-02-16 (Estimated); Results first posted 2019-10-30 (Actual); Last update posted 2019-11-15 (Actual); Status verified 2019-11

CONDITIONS: Diabetes; Peripheral Neuropathy; Pain
MeSH Terms: conditions — Diabetes Mellitus; Peripheral Nervous System Diseases; Pain | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Normal saline infusion then lidocaine infusion (Placebo Comparator): Intravenous infusion of normal saline over a 40 minute period. second intervention: Intravenous infusion of lidocaine [5mg/kg] over a 40 minute period.
  Interventions: Drug: lidocaine; Drug: Placebo
- Lidocaine infusion, then normal saline infusion (Active Comparator): Intravenous infusion of lidocaine [5mg/kg] over a 40 minute period. second intervention: Intravenous infusion of normal saline over a 40 minute period.
  Interventions: Drug: lidocaine; Drug: Placebo

INTERVENTIONS:
Drug: lidocaine — lidocaine is a sodium channel blocker/analgesic. It is approved for intravenous administration for cardiac arrhythmias.
Drug: Placebo — Normal saline, approved for hypovolemia, and homeostasis.

SUMMARY:
Diabetic nerve pain [painful diabetic peripheral neuropathy] is a common medical problem with few reliably effective treatments. There is some evidence that sensory testing may help determine how individuals will respond to analgesic therapy. In this study, the investigators are evaluating the relationship between sensory testing and subject response to lidocaine infusion therapy.

DETAILED DESCRIPTION:
Diabetic peripheral neuropathy [DPN] is caused by diabetes-related metabolic damage to the sensory nervous system. It affects more than 3 million Americans and is leading cause of nerve damage-associated pain worldwide. Currently approved drugs such as gabapentin, pregabalin, and duloxetine provide pain relief only in 1 out of 4 or 5 people with DPN, pointing to a great need to identify effective therapy for these patients. Recent literature suggests that certain methods of assessing sensory nerve function in neuropathic pain patients may provide prediction to individual analgesic response; however, no placebo-controlled studies have been performed with the primary goal of identifying treatment response predictors in DPN.

We propose in this study to examine whether sensory testing to determine mechanical pain threshold [MPT] or heat pain threshold [HPT] will predict the subject's response to IV lidocaine analgesic therapy. We hypothesize that people with painful DPN who have high MPT or HPT are more likely to respond to lidocaine treatment. This is a prospective, double blind, placebo-controlled study with the primary objective of determining whether the results from the sensory testing predict the response to systemic lidocaine in patients with painful DPN.

Consented subjects will attend a screening visit and two intervention visits, during which they will undergo sensory testing and receive intravenous lidocaine or placebo infusion in a cross-over design. At enrollment, each patient will be assigned a study number, which will match a previously prepared computer-generated list of randomization numbers to determine the sequence of interventions: lidocaine and then placebo, or vice versa. An unblinded research nurse coordinator will be assigned to match the study number with randomized treatment sequence, and this person will prepare the study medications, which will look identical. This research nurse coordinator will not be involved at any stage at patient assessment or data analysis. The participants and all other study personnel will be blinded to the treatment allocation.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18;
2. Diagnosis of Diabetes Mellitus (Fasting Plasma Glucose > 126 mg/dL and/or HbA1C >6.5%);
3. Distal symmetric pain in lower extremities with duration of more than 3 months;
4. Presence of either numbness or at least 1 sensory disturbance (increased or decreased sensitivity) in the feet.
5. Spontaneous pain with intensity of ≥ 4 on 0-10 Numerical Rating Scale (NRS).

Exclusion Criteria:

1. Not giving consent to participate in the study;
2. Unable to complete self-report pain questionnaire;
3. History of moderate to severe renal or liver failure;
4. History of other central or peripheral neurologic disorders;
5. History of cardiac arrhythmias;
6. Contraindication to intravenous lidocaine;
7. Pregnancy or lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2018-10-17 (Actual); Study Completion 2018-10-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Simon Haroutounian, PhD, Principal Investigator — Department of Anesthesiology, WUSTL
Locations (1):
- Washington University School of Medicine/Barnes Jewish Hospital, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One participant only received lidocaine infusion and did not return to receive saline infusion.
Groups:
- Saline First, Then Lidocaine: Intravenous infusion of normal saline (placebo) over a 40 minute period (Period 1). Intravenous infusion of lidocaine 5mg/kg IBW over a 40 min period (Period 2)
- Lidocaine First, Then Saline: Intravenous infusion of lidocaine 5mg/kg IBW over a 40 min period (Period 1). Intravenous infusion of normal saline (placebo) over a 40 minute period (Period 2).
Period: Period 1
Arm/Group | Saline First, Then Lidocaine | Lidocaine First, Then Saline
Started | 17 | 17
Completed | 17 | 17
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Saline First, Then Lidocaine | Lidocaine First, Then Saline
Started | 17 | 16 (One participant did not return for Period 2 treatment)
Completed | 17 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Saline First, Then Lidocaine | Lidocaine First, Then Saline | Total
Number analyzed (Participants) | 17 | 17 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (12) | 56 (10) | 57 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 16
  Male | 8 | 10 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 7 | 10
  White | 14 | 10 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 17 | 17 | 34
Average pain intensity within the past week [Median (Inter-Quartile Range); unit: units on a scale] — Average pain within the past week at study intake, assessed on a 0-10 Numerical Rating Scale, where 0 is no pain, and 10 is worst pain imaginable
  units on a scale | 6 [5 to 8] | 6.5 [5.5 to 7] | 6.25 [5 to 7.25]

OUTCOME MEASURES:

1. Primary Outcome: Change in Spontaneous Pain at 60-120 Minutes After Lidocaine Infusion Initiated (Assessed on 0-10 NRS)
Description: Spontaneous pain will be assessed on numerical rating scale NRS (0= no pain, 10=worst pain imaginable) prior to infusion and then repeatedly for 120 minutes. The outcome measure will use the average of pain intensity measured at timepoints in the 60-120 min range after beginning of infusion. The mean %change in pain (from baseline) will be compared between lidocaine and placebo arms.
Time Frame: Baseline compared to 60-120 minutes after starting the infusion
Population: Participants who completed both infusions and had non-zero pain scores at the start of each infusion.
Measure: Mean (Standard Deviation); unit: percentage of pain change from baseline
Groups:
- Normal Saline Infusion: Intravenous infusion of normal saline over a 40 minute period.
  Placebo: Normal saline, approved for hypovolemia, and homeostasis.
- Lidocaine Infusion: Intravenous infusion of lidocaine [5mg/kg] over a 40 minute period.
  lidocaine: lidocaine is a sodium channel blocker/analgesic. It is approved for intravenous administration for cardiac arrhythmias.
Arm/Group | Normal Saline Infusion | Lidocaine Infusion
Number analyzed (Participants) | 31 | 31
percentage of pain change from baseline | 33 (46) | 51 (40)
Statistical Analysis 1: Comparison: Normal Saline Infusion vs Lidocaine Infusion; Test type: Superiority; p = 0.03, t-test, 2 sided; Paired t-test

2. Secondary Outcome: Evoked Mechanical and Thermal Sensation at Baseline and 60 Minutes After Infusion Initiation.
Description: Thermal and mechanical responses will be assessed at baseline and 60 minutes after infusions. Evoked intensities measured on a 0-10 sensory scale, where 5 is normal sensation, a number lower than 5 is reduced sensation and a number higher than 5 is greater sensation.
Time Frame: - 60 minutes (baseline) and + 60 minutes of initiating infusion
Population: Participants who received both lidocaine and normal saline infusions were analyzed.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- Normal Saline: Prior to Infusion; Normal Saline: 60 Minutes After Infusion Initiation: Intravenous infusion of normal saline over a 40 minute period.
- Lidocaine: Prior to Infusion; Lidocaine: 60 Minutes After Infusion Initiation: Intravenous infusion of lidocaine [5mg/kg] over a 40 minute period.
Arm/Group | Normal Saline: Prior to Infusion | Normal Saline: 60 Minutes After Infusion Initiation | Lidocaine: Prior to Infusion | Lidocaine: 60 Minutes After Infusion Initiation
Number analyzed (Participants) | 33 | 33 | 33 | 33
score on a scale
  Cold intensity | 2 [1 to 4] | 4 [2 to 5] | 3 [1 to 4] | 3 [1 to 4]
  Heat intensity | 2 [0 to 3] | 2 [0 to 3.5] | 2 [0 to 3] | 1 [0 to 3]
  Brush intensity | 4 [3 to 5] | 4 [2 to 5] | 5 [2 to 5] | 4 [1.5 to 5]
  Pinprick intensity | 4 [1.5 to 6] | 3 [1 to 5.5] | 4 [1.5 to 6] | 3 [1 to 5.5]

3. Secondary Outcome: NPSI (Neuropathic Pain Symptom Inventory) Descriptors of Pain at Baseline and 60 Min After Infusion
Description: NPSI pain descriptors will be assessed prior to infusion of placebo and lidocaine (baseline) and again at 60 minutes post-infusion. Descriptors are expressed on a 0-10 scale; 0-minimum (least), and 10 maximum (worst) score.
Time Frame: Baseline to 60 minutes of initiating infusion
Population: Participants who received both lidocaine and normal saline infusions analyzed.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Normal Saline: Prior to Infusion | Normal Saline: 60 Minutes After Infusion Initiation | Lidocaine: Prior to Infusion | Lidocaine: 60 Minutes After Infusion Initiation
Number analyzed (Participants) | 33 | 33 | 33 | 33
score on a scale
  Does your pain feel like burning? | 3 [0 to 4] | 0 [0 to 2] | 3 [0 to 5] | 0 [0 to 1]
  Does your pain feel like squeezing? | 2 [0 to 3] | 0 [0 to 2] | 2 [0 to 4] | 0 [0 to 2]
  Does your pain feel like electric shocks? | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 3.5] | 0 [0 to 0]
  Does your pain feel like stabbing? | 0 [0 to 2] | 0 [0 to 0.5] | 0 [0 to 4.5] | 0 [0 to 0]
  Do you feel pins and needles? | 2 [0 to 5.5] | 0 [0 to 3.5] | 4 [0 to 5] | 0 [0 to 0]
  Do you feel tingling? | 3 [0 to 5] | 1 [0 to 3] | 4 [1.5 to 6] | 1 [0 to 3]

4. Secondary Outcome: Change in Spontaneous Pain Intensity as a Function of Baseline MPT
Description: Correlation between Mechanical Pain Threshold (MPT in mN) at baseline and reduction in spontaneous pain intensity (% reduction on 0-10 NRS) at 60-120 minutes (averaged) from the study drug infusion. The slopes (Pearson coefficients) of the correlation obtained from lidocaine vs. placebo will be compared.
Time Frame: baseline to 60-120 minutes after starting the infusion
Population: Participants who completed both infusions and had non-zero pain scores at the start of each infusion.
Measure: Number (95% Confidence Interval); unit: Pearson coefficient
Groups:
- Normal Saline Infusion: Intravenous infusion of normal saline over a 40 minute period.
- Lidocaine Infusion: Intravenous infusion of lidocaine [5mg/kg] over a 40 minute period.
Arm/Group | Normal Saline Infusion | Lidocaine Infusion
Number analyzed (Participants) | 31 | 31
Pearson coefficient | .249 [-.098 to .538] | .063 [-.308 to 0.404]

5. Secondary Outcome: Change in Spontaneous Pain Intensity as a Function of Baseline HPT
Description: Correlation between Heat Pain Threshold (HPT in degrees Celsius) at baseline and reduction in spontaneous pain intensity (% reduction on 0-10 NRS) at 60-120 minutes (averaged) from the study drug infusion. The slopes (Pearson coefficients) of the correlation obtained from lidocaine vs. placebo will be compared.
Time Frame: Baseline to 60-120 minutes after starting the infusion
Population: Participants who completed both infusions and had non-zero pain scores at the start of each infusion. Two additional participants excluded as they could not sense heat on test site.
Measure: Number (95% Confidence Interval); unit: Pearson coefficient
Arm/Group | Normal Saline Infusion | Lidocaine Infusion
Number analyzed (Participants) | 29 | 29
Pearson coefficient | .023 [-.372 to .493] | -.151 [-.467 to .206]

ADVERSE EVENTS:
Time Frame: 0-120 minutes after infusion initiation
Arm/Group | Normal Saline Infusion | Lidocaine Infusion
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/34
Other Adverse Events (participants affected / at risk) | 11/33 | 13/34
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Normal Saline Infusion (N=33) | Lidocaine Infusion (N=34)
Dry mouth (Skin and subcutaneous tissue disorders) | 8 | 13
Drowsiness (Nervous system disorders) | 4 | 9
Perioral numbness (Nervous system disorders) | 2 | 8
Dizziness (Nervous system disorders) | 1 | 6
Dysesthesia (Nervous system disorders) | 1 | 7
Nausea (Nervous system disorders) | 0 | 2
Blurred vision (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 1
Arrhythmia (Cardiac disorders) | 1 | 0
Slurred speech (Nervous system disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-24): https://cdn.clinicaltrials.gov/large-docs/03/NCT02363803/Prot_SAP_000.pdf